CLINICAL TRIAL: NCT00943982
Title: The Treatment of Uveitic Cystoid Macular Edema With Topical Interferon Gamma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090191; 09-EI-0191
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-24

CONDITIONS: Uveitis
Keywords: Cystoid Macular Edema; Intermediate Uveitis; Uveitis; OCT; Interferon-Gamma (IFN-Gamma)
MeSH Terms: conditions — Uveitis; Macular Edema; Uveitis, Intermediate | interventions — Interferon-gamma

INTERVENTIONS:
Drug: Interferon Gamma 1-b

SUMMARY:
Background:

* Uveitis is a serious inflammatory condition that affects the eye and can cause vision loss. A common secondary problem associated with uveitis is macular edema (swelling). The macula is the part of the eye that is important for central vision, and swelling of the macula can lead to further vision loss. This condition is usually treated by medicines that target the immune system, but these medicines sometimes do not work or may cause side effects.
* Interferon gamma-1b (Actimmune(Registered Trademark)) is a bioengineered protein that can alter the way inflammatory cells work in the immune system. Interferon gamma-1b is given as an intramuscular injection; however, this study will use the drug as an eye drop. This study represents the first time that interferon gamma-1b is given as an eye drop. Researchers hope that interferon gamma-1b will treat macular edema by decreasing the swelling in the back of the eye.

Objectives:

- To investigate the safety and effectiveness of treating uveitis-associated macular edema with interferon gamma-1b.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with macular edema associated with uveitis (in one or both eyes) for at least 3 months.

Design:

* Participants will have three planned clinic visits during this study over the course of 2 weeks.
* All participants will have a medical history and eye examination.
* When receiving the drops, participants will have optical coherence tomography (a detailed scan of the retina) 60 minutes and 30 minutes before the drops; upon receiving the drops; and 30, 60, and 120 minutes after receiving the drops.
* After receiving the drops, participants will have another eye examination, blood drawn for samples, and further scans.
* Participants will be asked to return to the NIH Clinical Center 1 week after receiving the drops for an evaluation....

DETAILED DESCRIPTION:
Objective: Information gathered from our laboratories suggests that cystoid macular edema (CME) is caused by the disequilibrium of the Jak/Stat and mTor signal transduction pathways in the retinal pigment epithelium (RPE). We wish to investigate whether stimulating the Jak/Stat pathway with topically applied interferon gamma-1b can be a therapeutic intervention for the treatment of CME secondary to uveitis. The objective of this study is to investigate the safety and tolerability of ocular instillations(s) of interferon gamma-1b as an effective treatment for CME secondary to uveitis.

Study Population: Five participants with CME secondary to intermediate, panuveitis or posterior uveitis will receive a topical ocular instillation(s) of interferon gamma-1b.

Design: This Phase I, non-randomized, prospective, uncontrolled, dose-escalation, single-center study will involve a one-time instillation or series of instillations of interferon gamma-1b on the cornea and measure the potential response with optical coherence tomography (OCT) . Treatment success is defined as a 25% decrease in excess central macular thickening at any timepoint post-instillation as compared to baseline. The first two participants will receive one instillation (each instillation contains 10 microg in 0.05 mL solution), the next two participants will receive two instillations and the final participant will receive three instillations. OCT will be obtained at -60 minutes, -30 minutes and just before the instillation(s). Repeat OCTs will be taken at +30 minutes, +60 minutes and +120 minutes and again at the end of the day. All participants will return for a one-week safety visit.

Outcome Measures: The primary outcome is the change in excess central macular thickening as measured by OCT in response to interferon gamma-1b as compared with baseline. Secondary efficacy outcomes include changes in macular volume as measured by OCT, visual acuity, intraocular pressure, and intraocular inflammation as graded upon slit lamp examination. Secondary safety outcomes include ocular surface irritation assessed by fluorescein staining of the cornea and conjunctiva to assess toxicity changes in subjective ocular pain assessments as compared to baseline, number and severity of systemic and ocular toxicities and adverse events and the proportion of participants with a visual loss of greater than or equal to 15 ETDRS letters.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant must be 18 years of age or older.
  2. Participant must understand and sign the protocol's informed consent document.
  3. Participant has a diagnosis of intermediate, panuveitis or posterior uveitis at least three months prior to study enrollment and has associated CME secondary to uveitis in at least one eye (the study eye).
  4. Participant has a central macular thickness greater than or equal to 250 microns in the study eye.
  5. Participant is willing to comply with the study procedures and is expected to be able to return for all study visits.
  6. Participant has visual acuity of 20/200 or better in the study eye.
  7. Female participants of childbearing potential must not be pregnant or breast-feeding.
  8. Both female participants of childbearing potential and male participants able to father a child must agree to practice an adequate contraception during the study and for six weeks following the administration of study medication. Acceptable methods of contraception include hormonal contraception (i.e. birth control pills, injected hormones dermal patch or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy).

EXCLUSION CRITERIA:

1. Participant is expected to be unable to tolerate the ocular instillation.
2. Participant is unable to undergo OCT testing.
3. Participant had herpes keratitis in the past.
4. Participant is diagnosed with multiple sclerosis.
5. Participant has a significant active infection (an infection requiring treatment as determined by the medical team) or a history of chronic or recurrent infections that in the principal investigator's best medical judgment would preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07-17; Primary Completion 2010-06-24 (Actual); Study Completion 2010-06-24 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in central macular thickness as measured by OCT as compared with baseline.

SECONDARY OUTCOMES:
Secondary outcomes include: changes in macular volume as measured by OCT, changes in visual acuity, changes in intraocular pressure and changes in intraocular inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrews HE, Nichols PP, Bates D, Turnbull DM. Mitochondrial dysfunction plays a key role in progressive axonal loss in Multiple Sclerosis. Med Hypotheses. 2005;64(4):669-77. doi: 10.1016/j.mehy.2004.09.001. PMID 15694681
- [Background] Artuch R, Aracil A, Mas A, Colome C, Rissech M, Monros E, Pineda M. Friedreich's ataxia: idebenone treatment in early stage patients. Neuropediatrics. 2002 Aug;33(4):190-3. doi: 10.1055/s-2002-34494. PMID 12368988
- [Background] Artuch R, Aracil A, Mas A, Monros E, Vilaseca MA, Pineda M. Cerebrospinal fluid concentrations of idebenone in Friedreich ataxia patients. Neuropediatrics. 2004 Apr;35(2):95-8. doi: 10.1055/s-2004-815830. PMID 15127307